CLINICAL TRIAL: NCT05198037
Title: Clinical Implications of FKBP5 in Post-stroke Neural Plasticity and Neuromodulation Effects
Brief Title: Clinical Implications of FKBP5 in Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021-02-002C
Record Dates: First submitted 2021-11-23; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Stroke
Keywords: Stroke; FKBP5; Motor; Transcranial direct current stimulation; Plasticity; Stress
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Anticipated 100 participants are assigned to the experimental or sham-controlled groups with an allocation rate of 1:1, for the clinical trial. In addition, another group of patients participates in the observational study (no intervention).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active transcranial direct current stimulation (tDCS) (Experimental): Weak direct currents with 2 mA are delivered 20 minutes per session (including 30s ramp-up and 30s ramp-down) during tailored upper extremity task practice. Total sessions are 20 over 10 days.
  Interventions: Device: Bihemispheric tDCS
- Sham tDCS (Sham Comparator): The device is automatically shut down after 2-minute stimulation. Treatment sessions and frequency are the same as the Experimental arm.
  Interventions: Device: Bihemispheric tDCS

INTERVENTIONS:
Device: Bihemispheric tDCS — The anode and cathode are placed over the ipsilesional and contralesional primary motor cortex (C3 or C4 based on 10-20 system), respectively. The size of the electrode is 5x5 cm.

SUMMARY:
With contemporary lifestyle changes and global aging, it is important yet unknown how stress interacts to post-stroke outcomes. This proposal aims to study the link between the stress-responsive FKBP51-related pathways and neural plasticity after stroke, elucidating FKBP5 gene polymorphisms and blood FKBP51 regulation in relation to brain excitability and functions, understanding the effects of transcranial direct current stimulation, and characterizing brain mechanisms for individualized early rehabilitation after stroke.

DETAILED DESCRIPTION:
Stress is an underestimated risk factor and also a consequence of cardiovascular diseases and stroke. FK506-binding protein 51 (FKBP51) modulates stress responses by acting as a co-chaperone that negatively regulates glucocorticoid receptor (GR) to cortisol binding and nuclear signaling. In an oxygen-glucose deprivation (OGD) model of acute mouse hippocampal slices, FKBP5 deletion reduced ischemic neuronal hyperexcitation, and cathodal electrical stimulation of OGD-injured wild-type decreased FKBP51 levels. However, clinical implications of FKBP5 polymorphisms and FKBP51 regulation in post-stroke outcomes and neuromodulation-induced plasticity are unknown. We aim to assess the link between FKBP5 polymorphisms and blood FKBP51 regulation after stroke, and their relationship with stroke phenotypes, brain connectivity and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ischemic or hemorrhagic stroke
* Aged 20-80 years old

Exclusion Criteria:

* FMA-UE is over 49 points
* Major psychiatric diseases
* Major neurologic diseases
* Global aphasia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of Upper Extremity, FMA-UE | Change score from baseline (~10 days poststroke) to 90 days poststroke
  Motor recovery of upper extremity poststroke

SECONDARY OUTCOMES:
Action Research Arm Test, ARAT | Change score from baseline (~10 days poststroke) to 90 days poststroke
  Motor function of upper extremity poststroke
Fugl-Meyer Assessment of Lower Extremity, FMA-LE | Change score from baseline (~10 days poststroke) to 90 days poststroke
  Motor recovery of lower extremity poststroke
Perceived Stress Scale-10 | Change score from baseline (~10 days poststroke) to 90 days poststroke
  Stress level poststroke
Protein and gene test | Change score from baseline (~10 days poststroke) to 90 days poststroke
  Protein expression poststroke and identifying genotypes of participants

OTHER OUTCOMES:
Resting-state structural and functional connectivity by magnetic resonance imaging | Change score from baseline (~10 days poststroke) to 90 days poststroke
  Connectivity-level plasticity post-intervention/poststroke

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan